CLINICAL TRIAL: NCT05782517
Title: I-gel Laryngeal Mask Versus Endotracheal Intubation for Laparoscopic Gynaecological Procedures (NoTube Study)
Brief Title: I-gel vs. Endotracheal Intubation for Laparoscopic Gynaecological Procedures
Acronym: NoTube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22228NoTube
Record Dates: First submitted 2022-12-21; First posted 2023-03-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2024-09

CONDITIONS: Intubation Complication; Laryngeal Mask Complication
Keywords: I-gel; Endotracheal Tube
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-gel (Experimental)
  Interventions: Device: Supraglottic Airway Device
- Endotracheal Tube (Active Comparator)
  Interventions: Device: Endotracheal Tube

INTERVENTIONS:
Device: Supraglottic Airway Device — Placement of an I-gel Supraglottic Airway Device.
  Other Names: I-gel; Laryngeal Mask
  Arms: I-gel
Device: Endotracheal Tube — Placement of an Endotracheal Tube.
  Other Names: Portex Tracheal Tube; ETT
  Arms: Endotracheal Tube

SUMMARY:
The goal of this interventional study is to compare the I-gel laryngeal mask, a type of supraglottic airway device (SGA), with endotracheal intubation in terms of safety, ease of use and adverse side effects for patients during gynecologic laparoscopic procedures at the Brussels Fertility Center in Brussels, Belgium.

DETAILED DESCRIPTION:
The NoTube study aims to compare an I-gel laryngeal mask with an endotracheal tube (ETT) during gynaecological keyhole surgery (laparoscopy) as part of a fertility trajectory.

Laparoscopy requires general anaesthesia. During this general anaesthesia, the airway is secured. Classically, this is done with an endotracheal tube. This is a hollow tube between the vocal cords (in the trachea) through which the anaesthetist can support the patient's breathing during the procedure. This procedure is also called intubation. A muscle relaxant is given to make the placement of an endotracheal tube easier. Placing an endotracheal tube during laparoscopic procedures is still considered the 'gold standard'. The lungs are protected from the aspiration of stomach contents. The principal risks of intubation are tissue damage (e.g., to the lips and trachea), sore throat and damage to tooth elements.

An alternative to an endotracheal tube is a laryngeal mask. A laryngeal mask is sometimes called a 'supraglottis device' because it is inserted above the vocal cords (glottis). A laryngeal mask is generally easier to insert, no muscle relaxation is required, and there is also less risk of sore throat and less chance of tooth damage. Since the laryngeal mask does not pass through the vocal cords, there is less protection against aspiration of stomach contents.

With the arrival of newer laryngeal masks (e.g. the I-gel laryngeal mask), they are increasingly used as an alternative to an endotracheal tube during short, laparoscopic procedures. From initial studies, a laryngeal mask appears to be as effective as an endotracheal tube, with fewer side effects, such as a sore throat. Initial investigations suggest no higher risk of aspiration of gastric contents. However, there are no studies yet comparing the use of an I-gel with an endotracheal tube during short laparoscopic procedures in the context of a fertility trajectory where the whole population (i.e., patients with a BMI higher than 35kg/m²) can participate in the study.

This study will assign patients to either the endotracheal or the I-gel group. The anaesthetic during the procedure is the same in the two groups. In the endotracheal group, an additional muscle relaxant will be given. After the procedure, the patient answers some questions about possible discomforts (e.g. sore throat, hoarseness...). The patient also completes a similar questionnaire on the first day after surgery. On day three after surgery, a study officer calls the patient to review some questions again. Finally, the patient receives a final questionnaire at the end of sick leave.

ELIGIBILITY:
Inclusion Criteria:

* The expected duration of the procedure does not exceed 2 hours
* Agreeing to participate in the study

Exclusion Criteria:

* The expected duration of the procedure is longer than 2 hours
* The patient suffers from restricted mouth opening, trismus, recent oral trauma or oral abscesses
* The patient has a BMI of more than 40 kg/m²
* The patient is known to have gastroparesis or another risk factor that would prevent you from being sober during the procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients of female biological sex are eligible for inclusion.
Enrollment: 120 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Leak fraction | Thirty seconds after placement of the airway device, 30 seconds after completing insufflation of the abdomen, 30 seconds after positioning the patient in 30° Trendelenburg, every 10 minutes Trendelenburg, and 30 seconds after closing the fascia.
  The leak fraction is defined as the leak volume divided by the inspired tidal volume. The leak volume is the difference between the inspired and expired tidal volumes.

SECONDARY OUTCOMES:
Number of attempts for placement of the airway device | Immediately after placement of the airway device.
  A maximum of three tries is attempted before converting to a different technique.
Total induction time | Immediately after completion of the first capnography square waveform.
  Time from when the palpebral reflex of the patient is abolished until the appearance of the first capnography square waveform.
Number of manipulations of the airway device | During surgery
  The number of times the anaesthesiologist manipulates the airway device to ensure adequate ventilation.
Blood staining on the airway device | Immediately after removing the airway device
  It is noted whether there is blood staining of the airway device.
The presence of nausea and vomiting | 30 minutes after removal of the airway device, 1 hour after removal and 2 hours after removal.
  Grading of nausea severity:
  * 0: No nausea
  * 1: Mild nausea, not requesting pharmacological rescue
  * 2: Moderate nausea, requesting pharmacological rescue
  * 3: Severe nausea resistant to pharmacological treatment
  Grading of Vomiting severity:
  * 0: No vomiting
  * 1: Mild Vomiting, not requesting pharmacological rescue
  * 2: Moderate vomiting, requesting pharmacological rescue
  * 3: Severe vomiting, resistant to pharmacological treatment
The presence of dysphagia | 30 minutes after removal of the airway device, 1 hour after removal and 2 hours after removal
  Presence of dysphagia:
  * 0: no dysphagia
  * 1: Mild, only rare episodes, not considered a significant problem
  * 2: Moderate, occasional difficulty swallowing specific foods (e.g. steak)
  * 3: Severe, frequent difficulties swallowing the majority of food
The presence of hoarseness | 30 minutes after removal of the airway device, 1 hour after removal and 2 hours after removal
  Presence of hoarseness:
  * 0: No hoarseness present
  * 1: Hoarseness noted by the patient
  * 2: Mild readily apparent hoarseness of voice
  * 3: Severe readily apparent hoarseness of voice
The presence of respiratory complications | 30 minutes after removal of the airway device, 1 hour after removal and 2 hours after removal
  * Grade 0: no respiratory complications
  * Grade 1: Any deviation from normal postoperative course without the need of pharmacological treatment or surgical, endoscopic and radiological intervention.
  * Grade 2: Requiring specific pharmacological treatment. For example, pneumonia requiring antibiotics.
  * Grade 3: Requiring surgical, endoscopic or radiological intervention.
  * Grade 4: Life-threatening condition requiring intensive care unit (ICU) admission
Overall satisfaction | Postoperative day one, day three and either day seven (for diagnostic laparoscopies) or day 14 (for all other surgeries).
  An online questionnaire completed by the patient. Pain intensity will be recorded using a visual analogue scale and measuring the distance between the 'no pain' point (0 millimeters) and the patient's mark. A longer distance equals more intense pain.
Quality of the surgical working conditions | During surgery
  The surgeon is asked every 10 minutes to asses the quality of the surgical conditions using the Leiden Surgical Rating Scale (L-SRS). The L-SRS is a Likert scale ranging from 1 to 5 where 1 indicates extremely poor conditions, 2 poor conditions, 3 acceptable conditions, 4, good conditions and 5 optimal conditions

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No